CLINICAL TRIAL: NCT07404722
Title: Urethral Plate Flap Versus Tunica Vaginalis Flap Corporoplasty for the Correction of Residual Severe Ventral Curvature After Urethral Plate Transection in Hypospadias Repair: A Single-Center, Randomized, Controlled, Non-Inferiority Study
Brief Title: Urethral Plate Flap vs. Tunica Vaginalis Flap for Residual Severe Ventral Curvature in Hypospadias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Wei Ru, Associate Chief Physician, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-IRB-0555-P-01
Record Dates: First submitted 2025-12-09; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Residual Severe Ventral Curvature; Transection of the Urethral Plate; Corporoplasty; Pedicled Tunica Vaginalis Flap (TVF); Novel Urethral Plate Flap (UPF); Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urethral Plate Flap Corporoplasty (Experimental): 1. After degloving and transecting the urethral plate, mobilize the urethral plate.
  2. Transect the tunica albuginea at the point of maximal curvature to fully correct the ventral curvature.
  3. Mobilize and open the tunica vaginalis sac, and harvest a pedicled Tunica Vaginalis Flap (TVF).
  4. Transfer the TVF to the ventral side to repair the tunica albuginea defect, and suture with 6-0 absorbable sutures.
  5. Mobilize the space between the scrotal skin and dartos fascia. Place 2 interrupted sutures between the external spermatic fascia near the testis and the dartos fascia at the scrotal base to fix the testis within the sub-dartos space.
  Interventions: Procedure: Urethral Plate Flap Corporoplasty
- Tunica Vaginalis Flap Corporoplasty (Active Comparator): 1. After degloving and transecting the urethral plate, mobilize the urethral plate.
  2. Transect the tunica albuginea at the point of maximal curvature to fully correct the ventral curvature.
  3. Mobilize and open the tunica vaginalis sac, and harvest a pedicled Tunica Vaginalis Flap (TVF).
  4. Transfer the TVF to the ventral side to repair the tunica albuginea defect, and suture with 6-0 absorbable sutures.
  5. Mobilize the space between the scrotal skin and dartos fascia. Place 2 interrupted sutures between the external spermatic fascia near the testis and the dartos fascia at the scrotal base to fix the testis within the sub-dartos space.
  Interventions: Procedure: Tunica Vaginalis Flap Corporoplasty

INTERVENTIONS:
Procedure: Urethral Plate Flap Corporoplasty — 1.After degloving and transecting the urethral plate, mobilize the urethral plate. 2.Transect the tunica albuginea at the point of maximal curvature to fully correct the ventral curvature. 3.Mobilize and open the tunica vaginalis sac, and harvest a pedicled Tunica Vaginalis Flap (TVF). 4.Transfer the TVF to the ventral side to repair the tunica albuginea defect, and suture with 6-0 absorbable sutures. 5.Mobilize the space between the scrotal skin and dartos fascia. Place 2 interrupted sutures between the external spermatic fascia near the testis and the dartos fascia at the scrotal base to fix the testis within the sub-dartos space.
  Arms: Urethral Plate Flap Corporoplasty
Procedure: Tunica Vaginalis Flap Corporoplasty — 1.After degloving and transecting the urethral plate, mobilize the urethral plate. 2.Transect the tunica albuginea at the point of maximal curvature to fully correct the ventral curvature. 3.Mobilize and open the tunica vaginalis sac, and harvest a pedicled Tunica Vaginalis Flap (TVF). 4.Transfer the TVF to the ventral side to repair the tunica albuginea defect, and suture with 6-0 absorbable sutures. 5.Mobilize the space between the scrotal skin and dartos fascia. Place 2 interrupted sutures between the external spermatic fascia near the testis and the dartos fascia at the scrotal base to fix the testis within the sub-dartos space.
  Arms: Tunica Vaginalis Flap Corporoplasty

SUMMARY:
The correction of ventral curvature in hypospadias follows a stepwise principle. Clinically, in some cases of hypospadias, residual severe ventral curvature (VC ≥ 30°) persists even after thorough skin degloving and transection of the urethral plate, due to the unbalanced development of the ventral and dorsal tunica albuginea of the corpus cavernosum. In such cases, ventral tunica albuginea incision and corporoplasty with a graft are mandatory.

Although the currently commonly used pedicled Tunica Vaginalis Flap (TVF) corporoplasty can effectively correct the curvature, it requires additional dissection of the scrotum and tunica vaginalis sac. This prolongs the operative time and poses risks of donor-site complications, such as testicular retraction and scrotal hematoma.

The novel Urethral Plate Flap (UPF) corporoplasty utilizes local pedicled urethral plate tissue for homologous repair. This study adopts a prospective, single-center, randomized, controlled, double-blind, non-inferiority trial design, enrolling 90 subjects. The aim is to verify that the therapeutic efficacy of the UPF technique in correcting such residual severe ventral curvature is non-inferior to that of TVF, while demonstrating significant advantages in surgical efficiency and donor-site safety.

This study aims, through a single-center, double-blind, RCT design, and under the strict indication of "residual severe ventral curvature after urethral plate transection," to verify efficacy via a "non-inferiority" hypothesis, and to verify safety and efficiency via a "superiority" hypothesis. The goal is to provide Level I evidence for the update of hypospadias guidelines, while simultaneously exploring the establishment of postoperative imaging evaluation standards.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months to 14 years.
* Diagnosis: Primary hypospadias (no history of prior hypospadias repair).
* Intraoperative Condition: Residual ventral curvature ≥ 30° confirmed by artificial erection test after transection of the urethral plate.
* Consent: Signed informed consent provided by the participant's legal guardian.

Exclusion Criteria:

① Glans diameter < 1 cm; ② Combined with cryptorchidism; ③ Combined with severe bleeding disorders or coagulation dysfunction.

Ages: 6 Months to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-02-22 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate of Ventral Curvature at 12 Months Postoperatively | 12 Months Postoperatively
  Recurrence of ventral curvature is defined as residual ventral curvature ≥ 10° on lateral photographs during artificial erection.

SECONDARY OUTCOMES:
Operative Time for Curvature Correction | Intraoperative
  Recorded as the time from the "incision of the tunica albuginea" to the "completion of tunica albuginea repair and confirmation of a straight penis" (in minutes). This metric specifically excludes the time taken for urethroplasty and penile skin reconstruction to minimize confounding factors.
Incidence of Donor-Site Complications | From enrollment to the end of treatment at 12 months
  Assessment of complications related to the graft harvest site, including:
  Testicular events: Postoperative testicular retraction/ascent (defined as the testis position being higher than the middle of the scrotum).
  Scrotal events: Scrotal hematoma, edema, and secondary infections caused by these conditions.
Continuity of the tunica albuginea | 12 months postoperatively
  Evaluation is performed by a sonographer blinded to group allocation using High-Frequency Penile Ultrasound Evaluation
  Evaluation Parameters:
  Continuity of the tunica albuginea (Categorized as: Continuous / Interrupted).
Echogenicity of the corpus cavernosum beneath the graft | 12 month postoperatively
  Evaluation is performed by a sonographer blinded to group allocation using High-Frequency Penile Ultrasound Evaluation Evaluation Parameters: Echogenicity of the corpus cavernosum beneath the graft (Assessed for consistency with the host cavernous tissue)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China